CLINICAL TRIAL: NCT02999347
Title: The PregnanT-study: Pregnancy Outcomes After TVT and Other Mid-urethral Sling (MUS) Procedures
Brief Title: Pregnancy After Tension-free Vaginal Tape and Other Mid-urethral Sling Procedures
Acronym: PregnanT
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ole Aleksander Jonsbu Dyrkorn, MD, Oslo University Hospital
Other Study IDs: 2015/434REK
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Urinary Incontinence; Urinary Stress Incontinence; Pregnancy Complications
Keywords: Treatment Outcome; Mid-urethral slings; Gynecologic Surgery Procedures
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Women having undergone at least one pregnancy/delivery after their MUS surgery
- Controls: Every case will be matched with two controls. The controls will be matched with the study cases' age and year of surgery (+- 2 years of age if a perfect match is not obtainable). These controls have not undergone a subsequent pregnancy/delivery.

SUMMARY:
The purpose of this study is to determine the interactions between pregnancy and urinary stress incontinence in women with a mid-urethral sling (MUS). The specific aims of the 2 sub studies are:

Study 1:

The main aims of Study 1 are to evaluate any potential impact on urinary stress continence after a pregnancy/delivery following MUS surgery, and to evaluate any potential differences in continence status based on the mode of delivery for these women.

Study 2:

The aim of Study 2 is to examine how obstetric factors may affect the degree of incontinence in women registered in The Norwegian female incontinence registry prior to surgical treatment. In addition, we want to explore if there are obstetric risk factors predicting failure of a MUS surgery performed after pregnancy/delivery.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is defined as involuntary leakage of urine on effort, or exertion, or on sneezing or coughing or laughing. This is the commonest form of incontinence in women affecting one in three over the age of 18 years with significant impact on their quality of life.

The Tension-free vaginal tape (TVT) was introduced in 1996 and has become one of the most widely used incontinence operations worldwide. In 2001, Delorme described a new mid-urethral sling using an outside-in transobturator approach, where the tape is inserted through the skin and the obturator foramen into the vagina (TOT). DeLeval developed a similar approach in 2003, where the tape is inserted inside-out from the vagina through the obturator foramen and the skin (TVT-O). TVT, TOT and TVT-O are collectively known as mid-urethral sling (MUS) operations.

Mid-urethral sling (MUS) operations can be performed as minimal invasive surgery in local anesthesia with short operative time and minimal surgical dissection. This type of surgery is now considered to be the standard surgical management for both SUI and mixed urinary incontinence (MUI) in which there is a predominant stress component. The short- and long term results are comparable to the Burch colposuspension and have been well documented.

Surgical treatment of SUI and MUI is generally recommended after the completion of childbearing for several reasons, one reason being that numerous studies have demonstrated pregnancy and delivery to be risk factors for SUI. Furthermore, in women treated with MUS, a new pregnancy and delivery might, in theory, change the position of the tape leading to the recurrence of incontinence symptoms. Women treated with MUS, who have recurrence of their SUI and MUI, also have a poorer outcome if given a second procedure (either a MUS or a bulking agent).

There is very limited knowledge about the consequences of a pregnancy in women who have undergone a mid-urethral sling operation, and only a few case reports exist in the literature. There is currently no consensus on either the management of a subsequent pregnancy or the mode of delivery after MUS surgery. Some clinical experts have claimed that vaginal delivery, where the baby's head exerts pressure on the anterior vaginal wall, may cause the tape to dislocate with potential injury to the bladder and urethra15. During the last decade, there has been a marked increase in the number of mid-urethral sling operations. This increase is probably due to the excellent short and long-term results, with less morbidity and a shorter hospital stay compared to colposuspension (the previous "gold standard" for SUI). It may therefore be expected in the future that more women of fertile age will request surgical treatment of SUI before the completion of their childbearing.

Several observational studies have shown that SUI is more prevalent in patients who have delivered at least one child. Obstetrical factors such as vaginal birth vs. elective cesarean section, parity, age at first pregnancy/birth and operative vaginal delivery have been associated with an increased risk of developing SUI. In addition, anal incontinence in fertile women is associated with SUI, probably due to more risk of pudendal nerve damage after an obstetrical anal sphincter injury with subsequent anal incontinence. Although obstetric factors are associated with the development of SUI, there are no studies on whether the same factors may negatively impact the outcome after SUI surgery.

The Norwegian Female Incontinence Registry (NFIR) was established in 1998. The purpose of the registry is to ensure the quality of incontinence surgery in Norway and that each department should be able to keep track of their results and use the information to improve the quality of their surgery. The majority of gynecological departments in Norway performing incontinence surgery report preoperative subjective and objective data, the type of incontinence procedures and complications, as well as 6-12 months' subjective and objective follow-up data to the registry. There are currently about 20 000 patients recorded in the registry, in a deidentified form, which means that only the Department that performed the operation has access to patient identity through a coded patient ID number (NFIR-number). Approximately 5 000 of these women are registered as being of childbearing age (< 45 years old) at the time of operation. In 2013 the NFIR obtained status as a National Quality Registry.

ELIGIBILITY:
Inclusion Criteria:

* Cases, consisting of women identified by the coupling of The Norwegian female incontinence registry and The medical birth registry of Norway as having undergone at least one pregnancy/delivery after their MUS surgery
* Controls, consisting of randomly selected women from Ullevål Hospital registered in the The Norwegian female incontinence registry with MUS surgery. Every case will be matched with two controls. The women will be matched with the study cases' age and year of surgery (+- 2 years of age if a perfect match is not obtainable). These controls have not undergone a subsequent pregnancy/delivery.

Exclusion Criteria:

* The only exclusion criterion will be the inability to give consent either due to reduced mental capacity or the lack of language skills in Norwegian or English.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women included in the Norwegian Female Incontinence Registry.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Subjective stress incontinence rates | Up to ten years
  Defined as the percentage of women having a stress incontinence index score < 5 on the validated questionnaire compared to women of equal age and follow-up time (also having undergone MUS surgery) not having undergone a subsequent delivery (controls)
Treatment satisfaction rate | Up to ten years
  Defined as the percentage of women stating "very satisfied" on the validated questionnaire in both cases and Controls.
The percentage of women not using urinary incontinence pads | Up to ten years
Any potential differences in subjective stress continence rates, the rate of women not using pads and treatment satisfaction rates based on the mode of delivery (spontaneous vaginal, operative vaginal and cesarean section) | Up to ten years

SECONDARY OUTCOMES:
Any potential adverse effects of undergoing a subsequent delivery after previous MUS surgery | Up to ten years
The continence status during pregnancy (before delivery) and whether any subjective incontinence was persistent or transient after delivery | Up to ten years
  Assesed on a validated questionnaire
The effect of time from MUS to subsequent delivery on stress continence status | Up to ten years
The impact on stress continence status from having undergone more than one subsequent delivery after MUS | Up to ten years
Differences in urgency score between controls and cases | Up to ten years
Any differences in subjective stress continence rates, treatment satisfaction rates or the rate of women not using pads when having undergone a subsequent delivery after previous MUS surgery based on the specific type of MUS (TVT, TOT or TVT-O) | Up to ten years
The effect of breastfeeding on subjective urinary stress continence rates having undergone pregnancy/delivery after MUS | Up to ten years

CONTACTS AND LOCATIONS:
Locations (1):
- Gynekologisk avdeling, Oslo Universitetssykehus Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided